CLINICAL TRIAL: NCT05986760
Title: Effects of Sports, Play and Active Recreation for Kids (SPARK) Versus Fundamental Motor Skill Training on Social and Motor Skills in Children With Autism Spectrum Disorder
Brief Title: Comparsion of SPARK and Fundamental Motor Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khadija liaquat (Other)
Responsible Party: Sponsor-Investigator, khadija liaquat, Senior lecturer, Riphah International University
Organization: Riphah International University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU-ASAD
Record Dates: First submitted 2023-06-15; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Motor Skill
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The SPARK is an evidence based plan designed to improve health-related well-being and to maintain the positive socialization and enjoyment of physical activities or academic achievements.(4) The SPARK discipline is in line with NASPE (National Association of Sport and PE) guidelines. A standard SPARK lesson will be delivered in two parts: a health fitness activity and a skill-fitness activity. In the health fitness activity part, there will be 13 activities that include aerobic dance, running games and jump ropes. In this part, the main focus will be on developing cardiovascular endurance and promotion by modifying the intensity, duration and complexity of the activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARK (Experimental): The SPARK is an evidence based plan designed to improve health-related well-being and to maintain the positive socialization and enjoyment of physical activities or academic achievements.(4) The SPARK discipline is in line with NASPE (National Association of Sport and PE) guidelines. A standard SPARK lesson will be delivered in two parts: a health fitness activity and a skill-fitness activity. In the health fitness activity part, there will be 13 activities that include aerobic dance, running games and jump ropes. In this part, the main focus will be on developing cardiovascular endurance and promotion by modifying the intensity, duration and complexity of the activities. The activities will be mostly aimed to develop abdominal and upper body strength.
  Interventions: Behavioral: SPARK
- Fundamental Motor training (Experimental): In terms of motor development, fundamental motor skills (FMS, e.g., locomotor and object manipulation)-such as running, jumping, throwing, and kicking-are considered the essential building blocks for further, more complex gross motor movement. (24) There will be 13 FMS activities including; running, jumping, Gallop, hopping, side gliding, skipping, leaping, catching, stationary dribbles, kicking, striking a stationary ball, overarm throw and underarm throw. FMS group will receive 30 sessions for 10 weeks (3 sessions per week, 60 min per session including CPT).
  Interventions: Behavioral: SPARK

INTERVENTIONS:
Behavioral: SPARK — Functional Motor training
  Other Names: FMS

SUMMARY:
It was a Randomized Clinical Trial.Data will be collected from Life care rehabilitation and special child facility.The study was completed within 6 months after approval of synopsis.The

calculated sample size, through WHO sample size calculator, using Bruininks- Oseretsky test's mean and standard deviation (Mean Dynamic Balance) as outcome

measure was 20 in each group. After adding 10% dropout the sample size will be 20+4=24 in each group; hence, overall sample size n= 20. Age range 5-12 years. Children with diagnosed Autism and age ranges between 5-12 will be included in the study.Convenient Sampling Technique was used to collect the data.There was two groups.In Group A SPARK therapy will be provided and in group 2 fundamental motor skill training will be provided. To assess the social skills Gilliam Autism Rating Scale-Second Edition (GARS-2) and for motor skills Bruininkse Oseretsky test of motor proficiency (BOTMP) was used.

DETAILED DESCRIPTION:
Autism Spectrum Disorder affects the social communication and fundamental motor skills of children. The current study will evaluate the effects of sports play and active recreation for kids (SPARK) versus fundamental motor skill training on social and motor skills in children with Autism spectrum disorder. It was a Randomized Clinical Trial.Data will be collected from Life care rehabilitation and special child facility.The study was completed within 6 months after approval of synopsis.The

calculated sample size, through WHO sample size calculator, using Bruininks- Oseretsky test's mean and standard deviation (Mean Dynamic Balance) as outcome

measure was 20 in each group. After adding 10% dropout the sample size will be 20+4=24 in each group; hence, overall sample size n= 20. Age range 5-12 years. Children with diagnosed Autism and age ranges between 5-12 will be included in the study.Convenient Sampling Technique was used to collect the data.There was two groups.In Group A SPARK therapy will be provided and in group 2 fundamental motor skill training will be provided. To assess the social skills Gilliam Autism Rating Scale-Second Edition (GARS-2) and for motor skills Bruininkse Oseretsky test of motor proficiency (BOTMP) was used. Analysis was carried out on SPSS version 27.

ELIGIBILITY:
Inclusion Criteria:

* Age range 5-9 years (11) • Diagnosed with an Autism Spectrum Disorder (ASD) based on Diagnostic and

Statistical Manual of Mental Disorders,

* Pervasive developmental disorder-not otherwise specified
* Asperger's disorder based on clinical judgment and supported by the Autism Diagnostic Observation Schedule
* Having moderate or greater behavioral problems as measured by a pretreatment score of >15 on the Aberrant Behavior Checklist-Irritability subscale
* Ability to follow directions and perform requested motor skill proficiency and executive function measures

Exclusion Criteria:

* Participants with diagnosed cognitive impairments

  * Unable to walk independently
  * History of traumatic injury
  * History of previous surgery history
  * Inability to understand the procedure and unwillingness to participate

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Social skills | Assessment took at 0 week of intervention and final reading was taken on 10th week of intervention
  Gilliam Autism Rating Scale-Second Edition (GARS-2)
Motor Skills: | Assessment took at 0 week of intervention and final reading was taken on 10th week of intervention
  Bruininkse Oseretsky test of motor proficiency (BOTMP)

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No